CLINICAL TRIAL: NCT05150236
Title: Phase II Study of Radionuclide 177Lu-PSMA Therapy Versus 177Lu-PSMA in Combination With Ipilimumab and Nivolumab for Men With MetastaticCastration Resistant Prostate Cancer (mCRPC)
Brief Title: EVOLUTION: 177Lu-PSMA Therapy Versus 177Lu-PSMA in Combination With Ipilimumab and Nivolumab for Men With mCRPC
Acronym: ANZUP2001
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other)
Collaborators: Prostate Cancer Foundation of Australia (Unknown); Bristol-Myers Squibb (Industry); Advanced Accelerator Applications (Industry); University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANZUP 2001
Record Dates: First submitted 2021-09-30; First posted 2021-12-09 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Prostate Cancer; Neoplasms by Site; Neoplasms; Prostatic Disease
MeSH Terms: conditions — Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Neoplasms by Site; Neoplasms; Prostatic Diseases | interventions — Pluvicto; Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination 177Lu-PSMA-617, Ipilimumab & Nivolumab (Experimental): 177Lu-PSMA (7.5GBq) given every 6 weeks up to 6 cycles in combination with concurrent ipilimumab (3mg/kg Q6W x 4 doses) and nivolumab (1mg/kg Q3W x 8 doses) followed by nivolumab monotherapy (480mg Q4W up to 18 doses) or until disease progression or unacceptable toxicity.
  Interventions: Drug: 177Lu-PSMA-617; Drug: Ipilimumab; Drug: Nivolumab
- 177Lu-PSMA-617 (Experimental): 177Lu-PSMA (7.5GBq) given every 6 weeks up to 6 cycles or until disease progression or unacceptable toxicity.
  Interventions: Drug: 177Lu-PSMA-617

INTERVENTIONS:
Drug: 177Lu-PSMA-617 — Patients will be given 7.5GBq of Lu-PSMA every 6 weeks up to 6 cycles unless there is unacceptable toxicity, commencing following result of 68Ga-PSMA PET within 28 days of registration.
  Other Names: 177Lutetium -PSMA 617 also referred to as 177Lu-PSMA
Drug: Ipilimumab — Patients will be given 3mg/kg of Ipilimumab every 6 weeks up to 4 doses unless there is unacceptable toxicity, concurrently with Lu-PSMA and Nivolumab.
  Other Names: YERVOY
  Arms: Combination 177Lu-PSMA-617, Ipilimumab & Nivolumab
Drug: Nivolumab — Patients will be given 1mg/kg of Nivolumab every 3 weeks up to 8 doses, concurrently with Lu-PSMA and Ipilimumab unless there is unacceptable toxicity. Followed by 480mg nivolumab monotherapy commencing at week 32. Nivolumab monotherapy will be given to patients every 4 weeks up to 18 doses, or until disease progression or unacceptable toxicity.
  Other Names: OPDIVO
  Arms: Combination 177Lu-PSMA-617, Ipilimumab & Nivolumab

SUMMARY:
This phase II study will investigate the activity and safety of radionuclide 177Lu-PSMA therapy versus 177Lu-PSMA in combination with Ipilimumab and Nivolumab in patients with metastatic castrate resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
This is an open label, randomised, stratified, multicentre phase 2 clinical trial recruiting 110 participants over 18 months and followed for 12 months. Participants will be randomised to 177Lu-PSMA in combination with Ipilimumab and Nivolumab and 177Lu-PSMA alone in a 2:1 ratio (using minimisation with a random component) stratified by prior exposure to docetaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older, with histologically confirmed adenocarcinoma of the prostate.
2. Castration-resistant metastatic prostate cancer (defined as disease progressing despite castration by orchidectomy or ongoing luteinising hormone-releasing hormone agonist or antagonist).
3. Patients must have progressed on prior novel AR targeted agents for treatment of prostate cancer. Progressive disease defined by at least one of the following:

   * PSA progression, minimum of two rising PSA values from a baseline measurement with an interval of ≥ 1 week between each measurement. The PSA value at screening should be ≥ 5ng/ml
   * Soft tissue or visceral disease progression as per RECIST 1.1
   * Bone progression: ≥ 2 new lesions on bone scan as per PCWG3
4. Target or non-target lesions according to RECIST 1.1 and PCWG3
5. Significant PSMA avidity on PET/CT using 68GaPSMA, defined as SUVmax ≥15 at a site of disease, and SUVmax ≥ 10 at other sites of disease ≥10mm (where there is no impact from partial voluming.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
7. Adequate bone marrow, hepatic and renal function documented within 28 days of registration, defined as:

   * Haemoglobin ≥90 g/L independent of transfusions (no red blood cell transfusion in last 4 weeks)
   * Absolute neutrophil count ≥1.5x109/L
   * Platelets ≥100 x109/L
   * Total bilirubin ≤1.5 x upper limit of normal (ULN) except for patients with known Gilbert's syndrome
   * Aspartate transaminase (AST/SGOT) and alanine transaminase (ALT/SGPT) ≤2.5 × ULN or ≤5 × ULN for participants with liver metastases
   * Serum creatinine ≤1.5 x ULN or a calculated creatinine clearance > 50mL/min (Cockcroft-Gault equation)
8. Patients must have a life expectancy ≥ 24 weeks.
9. Willing and able to comply with all study requirements, including treatment, timing and/or nature of required assessments
10. Signed, written informed consent.

Exclusion Criteria:

1. Prostate cancer with known significant sarcomatoid, spindle cell or neuroendocrine cell components, or metastasis of other cancers to the prostate.
2. 18F-FDG-PET/CT SUVmax ≥10 at a site of measurable disease with no concurrent PSMA expression > 10mm
3. Prior treatment with anti-PD1, anti-PD-L1/L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T cell co-stimulation or checkpoint pathways.
4. Patients must not have had more than one line of chemotherapy. If a patient has had docetaxel chemotherapy for hormone sensitive or castrate resistant setting, this will be considered one line.
5. Prior treatment with 177Lu-PSMA.
6. Patients with active, known, or suspected autoimmune disease. Sjogren's syndrome is considered an autoimmune disease. Exceptions: Patients with vitiligo, type I diabetes mellitus, residual hypothyroidism due to an autoimmune condition only requiring hormone replacement, or conditions not expected to recur in the absence of an external trigger, may be eligible.
7. Patients with a condition requiring systemic treatment with either corticosteroids (>10mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of registration. Inhaled or topical steroids, and adrenal replacement doses ≤ 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
8. Participants must have recovered from all AE due to previous therapies to ≤Grade 1 or baseline. Participants with ≤ Grade 2 neuropathy may be eligible.
9. Active malignancies within the previous 2-years with >30% probability of recurrence within 1 year. Melanoma in situ, basal cell or squamous cell carcinomas of skin, are permitted.
10. Significant infection, including chronic active hepatitis B, hepatitis C, or HIV. Testing for these is not mandatory unless clinically indicated.
11. Radiation or surgery within 2 weeks of randomisation.
12. Previous history of interstitial lung disease or non-infectious pneumonitis.
13. Administration of a live vaccine within 30 days prior to the first dose of study drug.
14. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
15. Inadequate contraception. Men must have been surgically sterilised or use a (double if required) barrier method of contraception.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
PSA progression free survival (PSA-PFS) at 1 year (PCWG3) | Date of randomisation to the date of first evidence of PSA progression at 53 weeks post randomisation.
  PSA progression is defined as a rise in PSA by ≥ 25% AND ≥ 2 ng/mL above the nadir (lowest PSA point). This needs to be confirmed by a repeat PSA performed at least 3 weeks later.

SECONDARY OUTCOMES:
PSA response rate (PSA-RR) | Date of randomisation through to study completion, approximately 3 years from start of recruitment. Early rises in PSA prior to 12 weeks will be disregarded in determining PSA response.
  PSA response rate is defined as the proportion of participants in each group with a PSA reduction of ≥ 50% from baseline.
Frequency and severity of adverse events (CTCAE v5.0) | Date of first dose of study treatment until 100 days after cessation of study treatment.
  CTCAE v5.0 will be used to measure frequency and severity of AEs during study treatment.
Radiological progression free survival (PCWG3/RECIST1.1) | Date of randomisation to the date of first evidence of progression on imaging (PCWG3 criteria for bone lesions and RECIST 1.1 for soft tissue lesions) assessed every 12 weeks through to study completion, approximately 3 years from start of recruitment.
  Radiographic PFS is defined as the interval from the date of randomisation to the date of first evidence of radiographic progression, or the date of last known follow-up without progression.
PSA progression free survival (PCWG3) | Date of randomisation through to study completion, approximately 3 years from start of recruitment.
  PSA progression free survival is defined as the interval from the date of randomisation to the date of first evidence of PSA progression or the date of last known follow-up without PSA progression.
Overall survival (OS) | Through to study completion, approximately 3 years from start of recruitment.
  OS is defined as the interval from the date of randomisation to date of death from any cause, or the date of last known follow-up alive.
Objective response rate (ORR) | Date of randomisation through to study completion, approximately 3 years from start of recruitment.
  ORR is defined as partial or complete response at any stage of the study (from the date of randomisation to date of subsequent anti-cancer treatment). RECIST 1.1 will be used to assess ORR in participants with measurable disease.
Duration of response | Date of randomisation through to first radiological progression or through to study completion, approximately 3 years from start of recruitment.
  Duration of response is defined as the interval from the date of first response (Complete Response / Partial Response as per RECIST 1.1) to the date of first documented radiological progression as per RECIST 1.1 in participants with measurable disease.
Time to treatment response | Date of randomisation through to study completion, approximately 3 years from start of recruitment.
  Time to treatment response is defined as the interval from the date of randomisation to the date of first response (Complete Response / Partial Response as per RECIST 1.1) in participants with measurable disease.
Aspects of Health Related Quality of Life (HRQoL) - 1 | Within 7 days prior to randomisation, assessed every 12 weeks, through to study completion, approximately 3 years from start of recruitment.
  The EORTC QLQ-C30 (European Organisation for Research on Treatment of Cancer - Quality of Life Questionnaire for cancer patients) instrument uses 28 questions about overall quality of life with each question answerable using a scale from 1 (not at all) to 4 (very much). Overall scores can be from a minimum of 28 indicating a better quality of life and higher scores with a maximum of 112 indicating lower overall quality of life. The questionnaire also has two summary questions which asks participants to rank 1) overall health and 2) overall quality of life on scale of from 1 (very poor) to 7 (excellent).
Aspects of Health Related Quality of Life (HRQoL) - 2 | Within 7 days prior to randomisation, assessed every 12 weeks, through to study completion, approximately 3 years from start of recruitment.
  Patient DATA Form (Patient Disease and Treatment Assessment Form - 47 items) is a simple, multi-item quality of life instrument based on 11-point numeric rating scales for a range of relevant symptoms and functions. It combines cancer specific items from the UBQ-C, GLQ-8 and LASA cancer-specific quality of life instruments.

OTHER OUTCOMES:
Association between Clinical Outcomes and Possible Prognostic/Predictive Biomarkers (tissue and circulating) including PBMCs, ctDNA and CTCs | Date of randomisation through to study completion, approximately 3 years from start of recruitment.
  Translational research will include identifying tissue and circulating biomarkers that are prognostic and/or predictive of response to treatment, safety and resistance to study treatment.
  These include but are not limited to analyses of:
  1. PBMC samples may be used for immunophenotyping or characterisation of the immune cell subsets in the periphery;
  2. ctDNA, immunological markers, and response data will be used to prospectively investigate the utility of early changes in ctDNA levels;
  3. CTCs may be enumerated and analysed for their potential to predict or correlate with toxicity and efficacy of immune checkpoint inhibitors.

CONTACTS AND LOCATIONS:
Overall Officials: Shahneen Sandhu, MBBS, FRACP, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (8):
- Australia (8):
  - St Vincents Hospital, Darlinghurst, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Royal Brisbane and Womens hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Sir Charles Gairdner, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Study protocol will be published in a peer-reviewed journal within 24 months.